CLINICAL TRIAL: NCT05544175
Title: NEUROMOdulation Pain Therapy in Combination With Intensive Physiotherapy on a Neurophysiological Basis Improves Not Only Pain But Also Mobility in Spastic Paraparesis
Brief Title: NEUROMOdulation Pain Therapy in Combination With Intensive Physiotherapy
Acronym: NEUROMOFY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kamila Řasová, assoc. prof. PhDr. Kamila Řasová, Ph.D., Charles University, Czech Republic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 092022
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Spinal Cord
Keywords: spinal cord stimulation; physiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NEUROMOdulation pain therapy in combination with intensive physiotherapy (Experimental): Neuromodulation therapy (low-voltage electrical stimulation of the posterior roots of the spinal cord) by electrodes inserted epidurally from a laminotomy in the lumbosacral region.
  Intensive, four hour per day, individual physiotherapy (soft techniques, methods based on neurophysiology, so-called neuroproprioceptive "facilitation, inhibition" (Vojta's reflex method, Motor programs activating therapy, Proprioceptive neuromuscular stimulation, Bobath concept) will be combined with methods of acquiring motor skills (individualized therapy using the knowledge of sensorimotor learning) will take minimally one month.
  Interventions: Procedure: NEUROMOdulation pain therapy in combination with intensive physiotherapy

INTERVENTIONS:
Procedure: NEUROMOdulation pain therapy in combination with intensive physiotherapy — Neuromodulation: Spinal cord stimulation affects nerve tissues with a defined electrical current. We will use low-voltage electrical stimulation of the posterior roots of the spinal cord in the MRI region of the localized conus medullaris. Electrodes are inserted epidurally from a laminotomy in the lumbosacral region.
  Physiotherapy will be based on recommendations for spinal patients.

SUMMARY:
In this project, the aim is to verify that neuromodulation therapy (spinal cord stimulation) in combination with intensive physiotherapy on a neurophysiological basis will lead to the restoration of mobility of lower limbs.

DETAILED DESCRIPTION:
So far, posterior spinal cord neurostimulation (NM SCS) has been applied as a standard in patients with the most severe forms of pharmacoresistant neuropathic pain. The most recent research of the last 1-2 years brings clinical findings that, in a mode and modified arrangement, it could even induce rhythmic muscle activity of the lower limbs and help in verticalization and assisted bipedal locomotion.

In this project, the aim is to verify that neuromodulation therapy SCS (spinal cord stimulation) in combination with intensive physiotherapy on a neurophysiological basis will lead to the restoration of mobility of lower limbs.

In the therapy, the neuronal circuits of the lumbosacral region, where the so-called central pattern generators for locomotion are located will be targeted. Neurostimulation of this area will generate motor movement patterns corresponding to the previous mapping of the corresponding muscle groups. These will be supported by intensive physiotherapy on a neurophysiological basis - thanks to it and the facilitation of movement by neurostimulation, global motor patterns will be triggered, and motor programs stored at the subcortical level will be activated. Their memorization and subsequent spontaneous retrieval will facilitate sensorimotor learning techniques.

Current research further shows that neurostimulation stimulates neurons in Rexed laminae 3-5, specifically a group of neurons designated as SC VSX2 and subsequently proprioceptive fibres. Physiotherapy will enhance the effect of neuromodulation by stimulating proprioceptors using soft and neurophysiologically based techniques. Proprioceptive fibres make connections to motoneurons and also ascend through the spinal cord to the brain, and thus reflex motor movements can be triggered. Information about them is carried to the brain by ascending pathways, and thus a free awareness of the movement facilitated by the neurostimulator occurs. All these mechanisms should potentiate plasticity (and lead to the restoration of locomotion.

ELIGIBILITY:
Inclusion Criteria:

spinal cord lesion

Exclusion Criteria:

other neurological conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle strength at 2 weeks, 6 weeks, 6 and 12 months | Pre-assessment (baseline testing), Post-assessment 1 (immediately after the end of two weeks hospitalisation), Post-assessment 2 (immediately after the end of one month hospitalisation), Follow up (6 and 12 month after beginning of the study).
  Hip flexion, abduction and extension, knee flexion and extension, plantar flexion and dorsiflexion using a microFET2 digital dynamometer. The higher value, the better function (higher strength).
Change in Spasticity at 2 weeks, 6 weeks, 6 and 12 months | Post-assessment 1 (immediately after the end of two weeks hospitalisation)
  Hip flexors, knee flexors and extensors, dorsal and plantar flexors using the Modified Ashworth scale. The higher value, the worse function (higher spasticity).
Change from Baseline Timed Up And Go at 2 weeks, 6 weeks, 6 and 12 months | Post-assessment 1 (immediately after the end of two weeks hospitalisation)
  The subject stands up from a chair, walks 3m, turns back, and sits down again as quickly and safely as possible while being timed. Higher times reflect worse mobility.
Change from Baseline Berg Balance Scale at 2 weeks, 6 weeks, 6 and 12 months | Post-assessment 1 (immediately after the end of two weeks hospitalisation)
  The subject stands up from a chair, walks 3m, turns back, and sits down again as quickly and safely as possible while being timed. Higher times reflect worse mobility.
Change from Baseline The 10 Metre Walk Test at 2 weeks, 6 weeks, 6 and 12 months | Post-assessment 1 (immediately after the end of two weeks hospitalisation)
  A performance measure used to assess walking speed in meters per second over 10 meters. Shorter times reflect better mobility.
Change from Baseline The 6 Minute Walk Test at 2 weeks, 6 weeks, 6 and 12 months | Post-assessment 1 (immediately after the end of two weeks hospitalisation)
  A long walking capacity test recording the maximal distance a subject walks at the fastest speed possible in 6 minutes. The more distance covered, the better the walking performance is.
Change in Walking Index for Spinal Cord Injury at 2 weeks, 6 weeks, 6 and 12 months | Pre-assessment (baseline testing), Post-assessment 1 (immediately after the end of two weeks hospitalisation), Post-assessment 2 (immediately after the end of one month hospitalisation), Follow up (6 and 12 month after beginning of the study).
  questionnaire from 0 to 20. Higher number means better function.

SECONDARY OUTCOMES:
Change in Visual Analogue Scale for pain at 2 weeks, 6 weeks, 6 and 12 months | Pre-assessment (baseline testing), Post-assessment 1 (immediately after the end of two weeks hospitalisation), Post-assessment 2 (immediately after the end of one month hospitalisation), Follow up (6 and 12 month after beginning of the study).
  scale from 0 to 10. Higher number means worse function (higher subjective feeling of pain)
Change in The Fatigue Scale for Motor and Cognitive Functions at 2 weeks, 6 weeks, 6 and 12 months | Pre-assessment (baseline testing), Post-assessment 1 (immediately after the end of two weeks hospitalisation), Post-assessment 2 (immediately after the end of one month hospitalisation), Follow up (6 and 12 month after beginning of the study).
  Questionnaire with 20 questions on fatigue. Higher number, worse fatigue.
Change in SYMBOL DIGIT MODALITIES TEST at 2 weeks, 6 weeks, 6 and 12 months | Pre-assessment (baseline testing), Post-assessment 1 (immediately after the end of two weeks hospitalisation), Post-assessment 2 (immediately after the end of one month hospitalisation), Follow up (6 and 12 month after beginning of the study).
  Cognitive testing (putting right symbols in 90 seconds). Higher number, better function.
Change in European Health Questionnaire at 2 weeks, 6 weeks, 6 and 12 months | Pre-assessment (baseline testing), Post-assessment 1 (immediately after the end of two weeks hospitalisation), Post-assessment 2 (immediately after the end of one month hospitalisation), Follow up (6 and 12 month after beginning of the study).
  questionnaire on Quality of Life. Higher value, better quality of life.
Change from Baseline World Health Organisation Disability Assessment Schedule 2.0 at 2 weeks, 6 weeks, 6 and 12 months | Pre-assessment (baseline testing), Post-assessment 1 (immediately after the end of two weeks hospitalisation), Post-assessment 2 (immediately after the end of one month hospitalisation), Follow up (6 and 12 month after beginning of the study).
  the 36-item questionnaire, higher score means higher disability
Change in the 36-Item Short Form Survey Instrument at 2 weeks, 6 weeks, 6 and 12 months | Pre-assessment (baseline testing), Post-assessment 1 (immediately after the end of two weeks hospitalisation), Post-assessment 2 (immediately after the end of one month hospitalisation), Follow up (6 and 12 month after beginning of the study).
  36 item questionnaire. Higher number, worse quality of life.
Change from Baseline Goal Attainment scale at 2 weeks, 6 weeks, 6 and 12 months | Pre-assessment (baseline testing), Post-assessment 1 (immediately after the end of two weeks hospitalisation), Post-assessment 2 (immediately after the end of one month hospitalisation), Follow up (6 and 12 month after beginning of the study).
  Each goal is rated on 5-point scale (-2 much less than expected, 0 achieved the expected level, 2 much more than expected). Higher score means a better outcome.
Change in the Spinal Cord Independence Measure at 2 weeks, 6 weeks, 6 and 12 months | Pre-assessment (baseline testing), Post-assessment 1 (immediately after the end of two weeks hospitalisation), Post-assessment 2 (immediately after the end of one month hospitalisation), Follow up (6 and 12 month after beginning of the study).
  17 item questionnaire. Higher number, better function (lower independence).

OTHER OUTCOMES:
Change from Baseline the serum level of Long non-coding ribonucleic acid (lncRNA) at 2 weeks, 6 weeks, 6 and 12 months | Pre-assessment (baseline testing), Post-assessment 1 (immediately after the end of two weeks hospitalisation), Post-assessment 2 (immediately after the end of one month hospitalisation), Follow up (6 and 12 month after beginning of the study).
  LncRNAs are defined as RNA transcripts >200 nucleotides with limited coding potential, but multiple function of binding different DNA, mRNAs and proteins, and they can be expressed under different conditions. As an improvement will be interpreted a significant mean fold change in gene expression (≥ 2.0, p value ≤ 0.05) between two groups following endogenous gene standardisation and normalization through control adjustment to a value of 1.0.
Change in pattern of brain activity at 6 and 12 months | Pre-assessment (baseline testing), Post-assessment 1 (immediately after the end of two weeks hospitalisation), Follow up (6 and 12 month after beginning of the study).
  fMRI will follow the changes in functional and structural brain connectivity. All fMRI examinations shall be performed in MR system Siemens Vida 3T located in IKEM using 64-channel RF head coil. Examination protocol will include not only essential structural imaging (3D SPACE FLAIR sequence with isotropic spatial resolution of 1 mm3), but also the measurement of functional connectivity using resting state fMRI and measurement of structural connectivity by means of the evaluation of spatial distribution of molecular diffusion (generalized DTI - diffusion tensor imaging, with 108 spatial directions and 3 b-factors allowing the reconstruction not only of fractional anisotropy but also the diffusion kurtosis imaging). The duration of the entire MR examination should not exceed 45 minutes. Extent activation, better value.
Change in muscle activity | Pre-assessment (baseline testing), Post-assessment 1 (immediately after the end of two weeks hospitalisation), Follow up (6 and 12 month after beginning of the study).
  Needle electromyography. Higher value, higher function.

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Řasová, assoc. prof., Principal Investigator — Department of rehabilitation, Third Faculty of Medicine, Charles University
Locations (1):
- Departmet of revmatology and rehabilitation, Faculty Thomayer Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
All data sharing terms and conditions and the nature of the relationship between the study and new user will be contained in a Data-sharing Agreement that will be issued and sighed before any data are handed out. The de-identification process for each patient is to ensure anonymization of individual patient's data, in order to be able to share IPD within the terms of participant's consent and ethics committee approval.
  The study policy on sharing defines the terms of privileged use by the study team. The research team requires to be appropriately notified and acknowledged in publications and other outputs of the transferred data (or analyses conducted by the study on the new users' behalf). The Data-sharing agreement will comprehend arrangements for data destruction or secure archiving.
  It is planned that the data will be placed into an online repository (to be specified later).
Supporting Information: Study Protocol, ICF
Time Frame: The IPD will be made available from 3-months months following the first publication of findings based on the data until 3 years following the first publication.
Access Criteria: The datasets will be prepared and might be reachable on a request. The study team formally reviews access requests for proposals. The data on an exclusive basis will be made available for third party use/ the new user, which can range from direct provision of data, data analysis collaboration, and/or scientific collaboration.
URL: http://ceros.mobi